CLINICAL TRIAL: NCT06560762
Title: A Phase 1, Open Label, Multiple Ascending Dose Study to Assess Safety and Tolerability of STM-01 in Participants With Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: Study in Participants With Heart Failure With Preserved Ejection Fraction (HFpEF)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Secretome Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Phase 1 STM-01 HFpEF Study
Record Dates: First submitted 2024-08-13; First posted 2024-08-19 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFpEF)

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, open-label, multi-center, dose-ranging study evaluating the safety and tolerability of STM-01 administered by intravenous infusion in participants with HFpEF. Up to 12 participants (2 cohorts) will be enrolled (Up to 6 participants, for 5 completers per cohort). Each successive cohort of participants will receive STM-01 at the following doses: 100.0 x 106 nMSCs, and 200.0 x 106 nMSCs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose arm (2 cohorts; 2 doses) (Other): Up to 12 participants will be enrolled (Up to 6 participants, for 5 completers per cohort). Each successive cohort of participants will receive STM-01 at the following doses: 100.0 x 106 nMSCs, and 200.0 x 106 nMSCs.
  Interventions: Drug: STM01

INTERVENTIONS:
Drug: STM01 — Neonatal mesenchymal stem cells (nMSCs),

SUMMARY:
A Phase 1, Open label, Multiple Ascending Dose Study to Assess Safety and Tolerability of STM-01 in Participants with Heart Failure with Preserved Ejection Fraction (HFpEF)

ELIGIBILITY:
Major Inclusion Criteria:

* Stable New York Heart Association (NYHA) Class II or III HF diagnosis, evident at least 6 months prior to enrolment as confirmed by medical history.
* Documented prior objective evidence of heart failure
* Screening ejection fraction ≥50%.
* Adequate bone marrow reserve and organ function at the Screening
* Receiving standard of care heart failure therapy at stable doses for at least 30 days prior to Screening.

Major Exclusion Criteria:

* Participant in any other study and has received any other investigational drug within 30 days prior to screening or 5-half-lives, whichever is longer, or any other investigational implanted device within 30 days prior to screening, or are taking part in a nonmedication study which, in the opinion of the Investigator, would interfere with study compliance or outcome assessments.
* Prior diagnosis of hypertrophic cardiomyopathy or a known infiltrative or storage disorder causing HFpEF and/or cardiac hypertrophy, such as amyloidosis, Fabry disease, or Noonan syndrome with LV hypertrophy.
* Persistent or permanent atrial fibrillation and is not therapeutically anticoagulated for at least the 4 weeks prior to the initial screening visit or is not adequately rate controlled within 6 months prior to informed consent according to investigator discretion.
* Other medical or psychiatric conditions that, in the opinion of the Investigator, would preclude obtaining voluntary consent/assent or would confound the objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Frequency, grade and relationship to STM-01 of unsolicited local and systemic AEs (any SAEs, MAAEs and AESIs ) during the 60-d follow-up period post IV infusion at D0 and D28 per the CTCAE v5.0 and clinical-safety laboratory parameters up to D 56. | Dose 1 (Day 0) till end of study (Day 56)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northwestern Medicine, Chicago, Illinois
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided